CLINICAL TRIAL: NCT05996055
Title: Comparison of the Benefits of Different Types of Wearable Respirator Support Devices for Critically Ill Patients in the ICU During Early Mobilization
Brief Title: A Comparative Study of Support Devices for Ventilator-Assisted ICU Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202303134DINA
Record Dates: First submitted 2023-07-31; First posted 2023-08-16 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Device Dislocation
Keywords: Intensive unit care; Early mobilization; Mechanical ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): initially using the Type A device (the NTUH version_support device)
  Interventions: Device: improved version_support device; Device: the NTUH version_support device
- experimental group (Experimental): initially using the Type B device (improved version_support device)
  Interventions: Device: improved version_support device; Device: the NTUH version_support device

INTERVENTIONS:
Device: improved version_support device — designed the NTUH version_support device based on the clinical suggestion.
  Other Names: type B support device
Device: the NTUH version_support device — original designed by NTUH
  Other Names: type A support device

SUMMARY:
Assisting critically ill patients with early mobilization or early ambulation during their stay in the intensive care unit (ICU) can reduce the duration of mechanical ventilation use, length of ICU or hospital stay, probability of complications during hospitalization, and sedation days in the ICU and improve disease prognosis. However, over 80% of critically ill patients have endotracheal tubes and require the use of mechanical ventilators in the ICU, and due to the numerous invasive treatments and tubes, there are high concerns regarding the safety of tube stability and risk of tube dislodgement during early mobilization. Although there are commercially available fixed tracheal tubes or external support devices for breathing tubes to prevent displacement, they do not solve the problems of the weight of the breathing tube during ambulation or endotracheal tube slippage. Therefore, through interdisciplinary collaboration, the investigator has designed a "wearable support device" (Type A support device). The unique design of the fixed frame uses a plug-in-latch shape to fix the Y-shaped breathing tube to the patient's chest position. In addition to reducing the displacement of the free section of the endotracheal tube downwards, it can also fix the main body of the breathing tube. The dual-disc strap method allows adjustment of the position and tightness for patients of different body sizes, and a single specification can be used for patients of various body shapes. Currently, a modified version of this wearable support device (Type B support device) has been designed based on clinical suggestions.The purpose of this study is to compare the feasibility, safety, and comfort of using the Type A-support device and the Type B-support device to assist in supporting breathing tubes during early ambulation in ICU patients using mechanical ventilators.

ELIGIBILITY:
Inclusion Criteria:

1. Glasgow Coma Scale score of ≥6,
2. relatively stable respiratory status (oxygen saturation >92%, settings on the mechanical ventilator: fraction of inspired oxygen ≤60%, positive end-expiratory pressure ≤10 cmH2O)
3. a stable cardiovascular system (resting heart rate ≤130 and >40 beats per minute)
4. no requirement for high-dose vasopressors >0.2 μg/kg/min).

Exclusion Criteria:

1. Patients with temporary limb immobilization as prescribed by the physician.
2. Patients with a tendency to bleed.
3. Patients with pre-existing mental abnormalities.
4. Patients who are expected to die within the next 24 hours or are primarily receiving palliative care in the intensive care unit.
5. Patients with sustained intracranial pressure elevation (> 20 millimeters of mercury (mmHg)).
6. Pregnant patients.
7. Uncontrolled epilepsy.
8. Acute myocardial infarction or rapidly progressing neuromuscular diseases occurring in the intensive care unit.
9. Patients with abnormal skin conditions such as skin abrasions, redness, swelling, etc., in the chest/back area.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
wearing time | From date of randomization up to 5 days
  the time taken to wear support device
removal time | From date of randomization up to 5 days
  the time taken to remove support device

SECONDARY OUTCOMES:
5-min heart rate variability (HRV) | From date of randomization up to 5 days
  including low-to-high-frequency power ratio (LF/HF) and standard deviation of NN intervals(SDNN)
mean values of the rapid shallow breathing index (RSBI) | From date of randomization up to 5 days
  recorded the ratio of respiratory rate (RR) and tidal volume (VT) and calulated by RR to VT
user self-reported function, and device satisfaction | From date of randomization up to 5 days
  self-made questionnaire
adverse event | From date of randomization up to 5 days
  Observe the abnormality of the skin on the chest/back of the base plate before and after wearing it; Record the number of incidents of accidental slippage of the external oral line while performing early ambulation while wearing the support device.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, Dr, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng, Taiwan

IPD SHARING:
Plan to Share IPD: No